CLINICAL TRIAL: NCT02097875
Title: A Phase 1 Dose Escalation/Expansion Study of BLZ-100 Administered by Intravenous Injection in Adult Subjects With Skin Cancer
Brief Title: Safety Study of a Fluorescent Marker to Visualize Cancer Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blaze Bioscience Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB-001; ACTRN12614000115639 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2014-03-25; First posted 2014-03-27 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Skin Neoplasms
Keywords: Skin cancer; Basal cell carcinoma; Squamous cell carcinoma; Melanoma
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Melanoma | interventions — tozuleristide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BLZ-100 (Experimental): A single dose of BLZ-100 (1, 3, 6, 12 or 18 mg) will be administered by intravenous injection approximately 48 hours prior to planned excision of skin tumor.
  Interventions: Drug: BLZ-100

INTERVENTIONS:
Drug: BLZ-100

SUMMARY:
Many types of cancer are primarily treated with surgery and patient survival is directly related to the extent to which the tumor is able to be removed. It is often difficult for surgeons to distinguish tumor tissue from normal tissue or to detect tumor cells that have spread from the original tumor site, resulting in incomplete removal of the tumor and reduced patient survival. In addition, in some sites, such as the brain, it is critical to avoid damage to normal tissue around the tumor to prevent adverse effects of surgery on function. We hypothesize that BLZ-100 will improve surgical outcomes by allowing surgeons to visualize the edges of the tumor and small groups of cancer cells that have spread to other sites in real-time, as they operate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age ≥ 18 years.
* Known or suspected non-metastatic basal cell or squamous cell carcinomas ≥10 mm longest diameter or non-metastatic melanoma ≥6 mm longest diameter scheduled for excision, without advanced disease.
* Written Informed Consent.
* Agree to the use of effective contraceptive from Baseline and for 30 days after treatment if either male or female of child bearing potential.
* Available for and able to comply with study requirements.

Exclusion Criteria:

* Women who are lactating/breastfeeding
* Women with a positive pregnancy test or who are planning to become pregnant during the duration of the study.
* Life expectancy <6 months.
* Karnofsky Performance Status of ≤70%.
* The following laboratory abnormalities:

  * Neutrophil count <1.5 x 10^9/L
  * Platelets <75 x 10^9/L
  * Haemoglobin <10 g/dL (may be determined following transfusion)
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2x upper limit of normal (ULN)
  * Total bilirubin >2x upper limit of reference range (unless Gilbert's syndrome or extrahepatic source as denoted by increased indirect bilirubin fraction)
  * International Normalized Ratio (INR) >1.5
  * Creatinine >1.5x ULN
* History of hypersensitivity or allergic reactions requiring corticosteroids, epinephrine and/or hospitalization.
* Uncontrolled asthma or asthma requiring oral corticosteroids.
* Clinically significant chronic inflammatory skin conditions, including psoriasis, atopic dermatitis and scleroderma, as determined by the investigator.
* Unstable angina, myocardial infarction, known or suspected transient ischemic events or stroke within 24 weeks of Screening.
* Uncontrolled hypertension.
* QTc (corrected QT interval) prolongation >450 msec.
* Receipt of photosensitising drugs within 30 days of screening.
* Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV).
* Any concurrent condition, including psychological and social situations, which, in the opinion of the investigator, would impact adversely on the subject or the interpretation of the study data.
* Known or suspected sensitivity to study product or excipients.
* Prior participation in this clinical trial (has received study product).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Within at least 1 week from baseline
  Safety will be assessed by physical examination and measurement of vital signs and laboratory safety parameters.

SECONDARY OUTCOMES:
Change in concentration of BLZ-100 in the blood | Prior to dosing and 1, 5, 15, 30, 60 and 90 minutes and 2, 3, 4, 6, 8, 12 and 24 hours post-dose
  BLZ-100 levels in blood will be analyzed by chemical means and these data will be used to calculate pharmacokinetic parameters.
Determination of a dose level for Phase 2 studies | At end of study - approximately 14 months

OTHER OUTCOMES:
Change in fluorescence signal in urine | Prior to dosing and at 0-4, 4-8, 8-12, 12-24 and 24-48 hours post-dose
  Fluorescence signal in urine samples will be measured using an infrared imaging system to determine the amount of BLZ-100 being excreted in the urine post-dosing.
Change in fluorescent signal in skin tumor and normal skin | Prior to dosing on day 1 and at 2, 4, 24 and 48 hours post-dose
  Fluorescence signal in skin tumor and normal skin will be measured in situ using the Fluobeam(TM) infrared imaging system.
Expression of biomarkers of response in excised skin tumor | 48 hours post-dose
  Immunohistochemistry will be used to measure the expression of other biomarkers of response, including Annexin A2, Ki67 and MMP2 (matrix metalloproteinase-2), in normal and tumor tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Spelman, MBBS FACD, Principal Investigator — Veracity Clinical Research Pty Ltd
Locations (1):
- Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland, Australia

REFERENCES:
- [Derived] Yamada M, Miller DM, Lowe M, Rowe C, Wood D, Soyer HP, Byrnes-Blake K, Parrish-Novak J, Ishak L, Olson JM, Brandt G, Griffin P, Spelman L, Prow TW. A first-in-human study of BLZ-100 (tozuleristide) demonstrates tolerability and safety in skin cancer patients. Contemp Clin Trials Commun. 2021 Aug 4;23:100830. doi: 10.1016/j.conctc.2021.100830. eCollection 2021 Sep. PMID 34401600